CLINICAL TRIAL: NCT07086378
Title: Evaluating the Efficiency and Tolerability of the Oxygenating Bite Block
Acronym: OBB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Robert Wong, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00003021
Record Dates: First submitted 2025-05-29; First posted 2025-07-25 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Endoscopy, Digestive System; Airway Anesthesia; Airway Control; Airway Management
Keywords: airway management; Upper endoscopy

STUDY DESIGN:
Intervention Model Description: Pilot study (ten subjects)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Oxygenating Bite Block (OBB) (Experimental): During the endoscopy procedure, the oxygenating bite block will be placed in the mouth instead of the standard and customary bite block.
  After the endoscopy procedure, the participant will be asked to complete a short questionnaire to find out their satisfaction with the level of sedation during the procedure, the tolerability of the device, and any discomfort.
  Interventions: Device: Oxygenating Bite Block

INTERVENTIONS:
Device: Oxygenating Bite Block — Oxygenating Bite Block will be used instead of the standard bite block.

SUMMARY:
This study will test an investigational bite block, which is a device placed inside the mouth to protect the teeth and used to keep the endoscope (a long, flexible tube that is placed down the throat and into the esophagus that contains a light and camera used to provide a visual of the area) in place. This Oxygenating bite block has been modified to allow the convenient use of an oral nasal cannula for administration of oxygen and sampling of end-tidal carbon dioxide (measurement of the amount of carbon dioxide exhaled at the end of a breath) during endoscopic procedures.

DETAILED DESCRIPTION:
This study will last one day and is completely voluntary.

The primary objective of this study is to evaluate the tolerability and efficacy of the device. The investigator will be testing how this device improves the flow of oxygen and provides safer sedation.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients scheduled to undergo upper endoscopy,
* Willingness and ability to sign an informed consent document,
* ASA class I - III obese adults,
* Subjects will be of diverse racial and ethnic backgrounds.

Exclusion Criteria:

* Patients deemed to be at significant airway risk,
* Under 18 years of age, since there is no justification to include them,
* Missing or loose incisor or canine teeth
* Temporomandibular joint disease
* Maxillofacial abnormalities (deformities of the jaw, lips, and tongue)
* Pregnant women, since there is no justification to include them,
* Emergency surgeries,
* Any other conditions that may interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wong, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
It is a small sample, only 10 subjects, it is a pilot study

REFERENCES:
- [Background] de Paulo GA, Martins FP, Macedo EP, Goncalves ME, Mourao CA, Ferrari AP. Sedation in gastrointestinal endoscopy: a prospective study comparing nonanesthesiologist-administered propofol and monitored anesthesia care. Endosc Int Open. 2015 Feb;3(1):E7-E13. doi: 10.1055/s-0034-1377835. Epub 2015 Jan 16. PMID 26134777
- [Background] Qadeer MA, Rocio Lopez A, Dumot JA, Vargo JJ. Risk factors for hypoxemia during ambulatory gastrointestinal endoscopy in ASA I-II patients. Dig Dis Sci. 2009 May;54(5):1035-40. doi: 10.1007/s10620-008-0452-2. Epub 2008 Nov 12. PMID 19003534

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxygenating Bite Block (OBB): During the endoscopy procedure, the OBB was placed in the mouth rather than the standard BB.
  After the endoscopy procedure, the participant will be asked to complete a short questionnaire to find out their satisfaction with the level of sedation during the procedure, the tolerability of the device, and any discomfort.
  OBB was used instead of the standard bite block.
Period: Overall Study
Arm/Group | Oxygenating Bite Block (OBB)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oxygenating Bite Block (OBB)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: OBB Device Feasibility
Description: SPO2 -Subject desaturation
Time Frame: During the upper endoscopy procedure
Population: SpO2 < 90%
Measure: Count of Participants; unit: Participants
Arm/Group | Oxygenating Bite Block (OBB)
Number analyzed (Participants) | 10
Participants | 3

2. Secondary Outcome: Tolerability of the Oxygenating Bite Block - Patients
Description: Questionnaire Satisfaction with the level of sedation and OBB tolerability?
Time Frame: After the endoscopy, up to 5 minutes
Population: All subjects (100%) expressed satisfaction with the level of sedation and OBB tolerability
Measure: Count of Participants; unit: Participants
Arm/Group | Oxygenating Bite Block (OBB)
Number analyzed (Participants) | 10
Participants | 10

3. Secondary Outcome: Tolerability of the Oxygenating Bite Block - Anesthesiologist
Description: Questionnaire Was the OBB easy to use, protected the subject's oral cavity, and oxygenated effectively?
Time Frame: After the endoscopy, up to 5 minutes
Population: Anesthesiologists expressed that the OBB was easy to use, protected the subject's oral cavity, and oxygenated effectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxygenating Bite Block (OBB)
Number analyzed (Participants) | 10
Participants | 10

4. Secondary Outcome: Tolerability of the Oxygenating Bite Block - Endoscopist
Description: Questionnaire - Endoscopist Did your patient tolerate the OBB well, and will you use it again?
Time Frame: After the endoscopy, up to 5 minutes
Population: Endoscopists expressed that the OBB was well tolerated and will you use it again.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxygenating Bite Block (OBB)
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 1 day (day of the procedure)
Description: Mortality was ZERO
Arm/Group | Oxygenating Bite Block (OBB)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT07086378/Prot_SAP_000.pdf
  • Study Protocol and Informed Consent Form (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT07086378/Prot_ICF_001.pdf